CLINICAL TRIAL: NCT02188966
Title: Telemedical Solutions in Medical Emergencies, Advantages and Disadvantages for Patients, Healthcare Professionals, and Healthcare System. Study 4: Application of Geographical Information System Data in the Emergency Department, Effect on Trauma Team and Medical Emergency Team Wait - a Before and After Study
Brief Title: Application of Geographical Information System Data in the Emergency Department, Effect on Trauma Team and Medical Emergency Team Wait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Horsens (Other); Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NRAA4
Record Dates: First submitted 2014-05-12; First posted 2014-07-14 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2014-03

CONDITIONS: All Acutely Ill or Injured Patients
Keywords: Geographic Information System; Emergency Care Information Systems; Telemedicine; Emergency Hospital Service
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Geographical Information System (Experimental): Availability of Geographical Information System data from ambulances destined for the Emergency Department of Regional Hospital Horsens.
  Interventions: Device: Geographic Information System

INTERVENTIONS:
Device: Geographic Information System — GIS data is delivered by "SimaTech Enterprise System" communicating via the mobile network and TETRA (in Denmark called SINE). It is developed as a Java Enterprise application and is executed on a JBOSS application platform
  Other Names: "ADO - AMK Dynamisk Overvågning" (Emergency Medical Dispatch Dynamic Surveillance)

SUMMARY:
In the Emergency Department Regional Hospital Horsens a monitor will display Geographical Information System data (GIS data) for all ambulances with the hospital as final destination. The location, estimated time of arrival (ETA) and urgency code for the ambulances will be showed. Furthermore the patient's name, personal identification number and the primary message received by the emergency medical dispatch center resulting in ambulance dispatch will be displayed. This may enable the coordinating nurse to optimize timing of the ad hoc trauma team and medical emergency team activation. The teams are activated if the patient's condition is assessed to be of the highest urgency and/or severity - triage 1 or "red". The coordinating nurse makes this assessment on the basis of information from the ambulance personnel and makes the decision to activate the team and when to do it. In this study the investigators want to examine if the availability of GIS data in the emergency department results in reduced waiting time for the members of the trauma team and medical emergency team. The study will be conducted as a before and after study.

ELIGIBILITY:
Inclusion Criteria:

* Critically Ill or Severely injured patients transported by ambulance
* Patients must be in triage category 1/"red"
* Emergency Medical Team og Trauma Team must be activated.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Waiting time | Time from activation of trauma team to arrival of patient, expected assesment within 1 minute after patients arrival, expected to be presented up to 36 months after assesment .
  Triage 1 or "red" of a patient indicates the highest urgency and/or severity of illness. If the coordinating nurse at the emergency department assess that a patient on the to the department is "red" the trauma team or medical emergency team is activated. The time is registered automatically in the internal telephone system of the hospital. The patient's time of arrival is registered manually. The time from activation to arrival can then be calculated and is defined as "Waiting time".

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Raaber, MD, Principal Investigator — Central Denmark Region; Erika Christensen, MD, medical director, Study Director — Central Denmark Region
Locations (1):
- Emergency Departmartment Regional Hospital Horsens, Horsens, Central Denmark Regione, Denmark

REFERENCES:
- [Derived] Raaber N, Duvald I, Riddervold I, Christensen EF, Kirkegaard H. Geographic information system data from ambulances applied in the emergency department: effects on patient reception. Scand J Trauma Resusc Emerg Med. 2016 Mar 31;24:39. doi: 10.1186/s13049-016-0232-5. PMID 27029399